CLINICAL TRIAL: NCT00764972
Title: A Phase IB/II Trial of Combination of Vinorelbine With Sorafenib (BAY 43-9006) as First-Line Treatment in Patients With Metastatic Breast Cancer
Brief Title: Phase IB/II Trial Combining Vinorelbine With Sorafenib as First-Line Treatment in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Cristina Attard, BSc Oncology Project Specialist, Bayer HealthCare Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McG 0713
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Metastatic Breast Cancer
Keywords: To evaluate the use of sorafenib added to vinorelbine chemotherapy, to find out which are the doses of two drugs can be safely combined
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and Vinorelbine (Experimental)
  Interventions: Drug: Sorafenib and Vinorelbine

INTERVENTIONS:
Drug: Sorafenib and Vinorelbine — vinorelbine, administered as a brief infusion twice every three weeks (on day 1 and 8 of 21-day cycles);
  sorafenib, that you will take orally every day, at the dosage that your study doctor will prescribe.
  Other Names: BAY 43-9006

SUMMARY:
This is a phase IB/II trial of sorafenib, a new tyrosine kinase inhibition of multiple genes that is active against renal cancer, plus vinorelbine, a chemotherapy agent active in breast cancer.

The investigators are combining these 2 drugs in order to determine if the investigators can increase the activity of vinorelbine in metastatic breast cancer patients.

Patients with measurable metastatic breast cancer without previous chemotherapy for metastatic disease are eligible for the protocol. They will be treated with 2 different dose levels of sorafenib in order to determine the most tolerable dose.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by histologically proven metastatic breast cancer.
* Tumor not susceptible to therapy with trastuzumab, defined as FISH negative for HER-2 amplification or immunohistochemistry 0-1+ for HER-2 expression.
* Female, age ≥ 18.
* Documented measurable disease by appropriate radiologic imaging according to RECIST criteria (see Appendix E). Lesions in previously irradiated areas are not considered measurable disease, unless progression has been documented post-radiation.
* ECOG performance status 0-1 (see Appendix B)
* Life expectancy > 6 months.
* Adequate bone marrow function, as indicated by:

  * Hemoglobin ≥ 90 g/L
  * Neutrophils ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
* Adequate renal function, as indicated by serum creatinine ≤1.5 times the upper limit of normal and/or Creatinine Clearance calculated as >50% lower normal limit, or estimated as ≥ 50 ml/min (Appendix C).
* Adequate liver function, as indicated by:

  * bilirubin ≤ 1.5 times upper normal limit;
  * AST and ALT ≤ 2 times upper normal limit.
* Left ventricular ejection fraction (LVEF) ≥50% as measured by either multigated acquisition (MUGA) scan or echocardiogram (ECHO).
* No therapy for breast cancer in the 4 weeks preceding the therapy start.
* Women of childbearing potential must be using adequate contraception and have a negative pregnancy test at the time of enrollment.
* Patient able to understand and give written informed consent.

Exclusion Criteria:

* Patients with locally advanced breast cancer or stage IIIb only.
* Presence of only non-measurable disease.
* Previous (neo)adjuvant chemotherapy with vinorelbine.
* Any previous anti-angiogenic therapy.
* Any previous chemotherapy for metastatic breast cancer. Previous hormonal treatments or radiotherapy for metastatic disease are allowed.
* Radiotherapy, chemotherapy or hormonal therapy for breast cancer in the last 4 weeks prior to starting the study treatment.
* Major surgery within 4 weeks of first study treatment, or minor surgery (including placement of an access device) within 7 days of therapy start.
* Presence of life-threatening disease or central nervous system localizations.
* Evidence of HER-2 positive breast cancer, defined as FISH-positive for amplification or score 3+ by immunohistochemistry.
* Any other possibly active primary tumor, except basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Clinically significant hepatic disease with respect to hepatitis B, hepatitis C, cirrhosis or other liver diseases.
* Uncontrolled bacterial, viral or fungal infection.
* Previous history of ischemic disease.
* Patients with previous history of thrombo-embolic events, or with documented risk factors for thrombotic disease other than cancer.
* History of gross hemorrhage within the past 6 months (e.g., hemoptysis or hematuria requiring medical intervention).
* Uncontrolled hypertension.
* Other serious medical conditions, such as uncontrolled cardiac disease, severe pulmonary disease, uncontrolled diabetes.
* Patient exhibiting confusion or disorientation.
* Any condition (medical, social, psychological, geographical) that would prevent adequate follow-up.
* Patient is pregnant, or is breast-feeding, or is unwilling to use adequate contraception.
* Failure to give informed consent.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Confirmed complete response (CR) or partial response (PR), defined according to RECIST criteria, persisting 4 weeks after the initial documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Panasci, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ferrario C, Strepponi I, Esfahani K, Charamis H, Langleben A, Scarpi E, Nanni O, Miller WH Jr, Panasci LC. Phase I/II Trial of Sorafenib in Combination with Vinorelbine as First-Line Chemotherapy for Metastatic Breast Cancer. PLoS One. 2016 Dec 19;11(12):e0167906. doi: 10.1371/journal.pone.0167906. eCollection 2016. PMID 27992451